CLINICAL TRIAL: NCT01691781
Title: The Renin-Angiotensin-Aldosterone System and Parathyroid Hormone Control: The RAAS-PARC Study
Acronym: RAAS-PARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anand Vaidya, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012p0001961
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Hyperparathyroidism
Keywords: Hyperparathyroidism; Renin-angiotensin-aldosterone system; ACE inhibitors
MeSH Terms: conditions — Hyperparathyroidism | interventions — Lisinopril

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lisinopril (Experimental): Lisinopril - open-label, 2.5-40mg daily
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Lisinopril — Each subject will receive one week of lisinopril and return for repeat for blood measurements.

SUMMARY:
This study will evaluate whether commonly used blood pressure medications called "ACE inhibitors" can lower parathyroid hormone.

DETAILED DESCRIPTION:
The RAAS-PARC study will evaluate whether angiotensin-converting enzyme inhibitors (ACEi) can lower parathyroid hormone (PTH) in normal controls and in individuals have a diagnosis of primary hyperparathyroidism.

Emerging data has implicated the renin-angiotensin-aldosterone system (RAAS) activity with increased PTH. The principal investigator, and other investigators, have previously shown that inhibiting the RAAS may lower PTH. The current study will focus on:

1. Normal Physiology: Does an ACEi (which lowers angiotensin II and aldosterone) reduce PTH in normal individuals?
2. Pathophysiology: Does an ACEi reduce PTH in individuals with primary hyperparathyroidism?

The results of this study may have important implications for cardiovascular and skeletal health, as both the RAAS and PTH have been implicated as mediators of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with with no medical problems (n=15) and individuals with primary hyperparathyroidism (n=30)
* normal blood pressure or stage 1 hypertension that is either untreated, or adequately treated with a single anti-hypertensive medication.
* Age >18 years and <80 years
* Estimated GFR > 60ml/min

Exclusion Criteria:

* Chronic Kidney Disease or eGFR<60
* Stage 2 or Stage 3 hypertension or the use of more than 1 antihypertensive drug
* Type 2 Diabetes Mellitus that is not controlled by diet or Metformin alone or with a Hemoglobin A1c >7.5%
* History of liver failure
* History of heart failure
* The use of typical or atypical antipsychotic medications or lithium.
* Chronic inflammatory conditions (such as inflammatory bowel disease or arthritis) that are treated with prescribed doses of NSAIDs or glucocorticoids
* The use of prescribed doses of potassium supplements.
* Illness requiring overnight hospitalization in the past 6 months
* Active tobacco or recreational drug use
* Pregnancy or current breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Vaidya, MD, MMSc, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zaheer S, Brown JM, Connors M, Williams JS, Adler GK, Vaidya A. Angiotensin-Converting Enzyme Inhibition and Parathyroid Hormone Secretion. Int J Endocrinol. 2017;2017:4138783. doi: 10.1155/2017/4138783. Epub 2017 Jul 20. PMID 28808443

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants had to undergo a washout of ACE inhibitors (if applicable) during which time their blood pressure had to remain within safety parameters, and they had to complete a controlled sodium diet.
Groups:
- Primary Hyperparathyroidism: Participants with Primary Hyperparathyroidism enrolled to receive open label lisinopril.
- Normal: Participants without primary hyperparathyroidism enrolled to receive open label lisinopril.
Period: Overall Study
Arm/Group | Primary Hyperparathyroidism | Normal
Started | 19 | 22
Completed | 12 | 15
Not Completed | 7 | 7
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Normals: Participants without primary hyperparathyroidism enrolled to receive open label lisinopril.
- Total: Total of all reporting groups
Arm/Group | Primary Hyperparathyroidism | Normals | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (15.6) | 39.6 (12.7) | 44.9 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 15 | 27
Parathyroid Hormone at Baseline [Mean (Standard Deviation); unit: pg/mL] | 79.5 (21.6) | 33.3 (25.4) | 53.8 (33.0)
Serum calcium [Mean (Standard Deviation); unit: mg/dL] | 10.6 (0.5) | 9.4 (0.4) | 9.9 (0.7)
Urinary Aldosterone Excretion Rate at baseline [Mean (Standard Deviation); unit: mcg/24 hours] | 11.7 (18.3) | 5.7 (3.5) | 8.2 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Parathyroid Hormone Following 1 Week of ACE Inhibitor Administration
Description: PTH values 1 week following ACE inhibitor therapy
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Primary Hyperparathyroidism | Normal
Number analyzed (Participants) | 12 | 15
pg/mL | 70.9 (19.6) | 32.5 (16.7)
Statistical Analysis 1: Comparison: Primary Hyperparathyroidism; The statistical analysis compared the change in PTH, before and after ACE inhibitor therapy, among participants with primary hyperparathyroidism; Test type: Superiority; p = 0.049, t-test, 2 sided — This p-value reflects the difference in PTH means among participants with primary hyperparathyroidism
Statistical Analysis 2: Comparison: Normal; The statistical analysis compared the change in PTH, before and after ACE inhibitor therapy, among normal control participants (without primary hyperparathyroidism); Test type: Superiority; p = 0.80, t-test, 2 sided — This p-value reflects the difference in PTH means among normal control participants without primary hyperparathyroidism

2. Secondary Outcome: Urinary Aldosterone Excretion Measurements Following 1 Week of ACE Inhibitor Therapy
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mcg/24 hours
Arm/Group | Primary Hyperparathyroidism | Normal
Number analyzed (Participants) | 12 | 15
mcg/24 hours | 7.8 (8.9) | 6.1 (9.1)
Statistical Analysis 1: Comparison: Primary Hyperparathyroidism; The statistical analysis compared the change in urinary aldosterone excretion rate, before and after ACE inhibitor therapy, among participants with primary hyperparathyroidism; Test type: Superiority; p = 0.22, t-test, 2 sided — This p-value reflects the comparison of means among the primary hyperparathyroidism group only
Statistical Analysis 2: Comparison: Normal; The statistical analysis compared the change in urinary aldosterone excretion rate, before and after ACE inhibitor therapy, among normal control participants without primary hyperparathyroidism; Test type: Superiority; p = 0.86, t-test, 2 sided — This p-value reflects the mean difference in 24h aldosterone excretion rate among normal control participants without primary hyperparathyroidism

3. Secondary Outcome: Serum Calcium Following 1 Week of ACE Inhibitor Administration
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Primary Hyperparathyroidism | Normal
Number analyzed (Participants) | 12 | 15
mg/dL | 10.5 (0.4) | 9.5 (0.3)
Statistical Analysis 1: Comparison: Primary Hyperparathyroidism; The statistical analysis compared the change in serum calcium, before and after ACE inhibitor therapy, among participants with primary hyperparathyroidism; Test type: Superiority; p = 0.48, t-test, 2 sided — This p-value reflects the statistic for the comparison of mean calcium levels for the primary hyperparathyroidism group
Statistical Analysis 2: Comparison: Normal; The statistical analysis compared the change in serum calcium, before and after ACE inhibitor therapy, among normal control participants without primary hyperparathyroidism; Test type: Superiority; p = 0.80, t-test, 2 sided — This p-value reflects the statistic for the comparison of mean calcium levels for the normal control participants without primary hyperparathyroidism

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Primary Hyperparathyroidism | Normal
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 2/12 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Hyperparathyroidism (N=12) | Normal (N=15)
Weakness (General disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This a small physiology pilot study that is open-label and non-randomized. The intervention was an ACE inhibitor, an approved therapy. Results have physiologic implications, but treatment implications are not intended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No